CLINICAL TRIAL: NCT05993572
Title: Does Healthy Aging Team-supported Home-care Services Pilot Program Reduce ED Visits? A Prospective before-and After-intervention Study
Brief Title: HEalthy Aging Team Supported Home-care Services (HEAT-YASAM)
Acronym: HEAT-YASAM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Gulhane Training and Research Hospital (Other Government)
Collaborators: Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Bilal Katipoglu, Associate Professor, Gulhane Training and Research Hospital
Other Study IDs: 2023-3-24
Record Dates: First submitted 2023-07-21; First posted 2023-08-15 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Frailty; Dementia; Depression; Malnutrition; Old Age; Debility; Drug Use
MeSH Terms: conditions — Frailty; Dementia; Depression; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Comprehensive Geriatric Assessment — Comprehensive Geriatric Assessments include functional status, fraility comorbidity, cognition, mental health, social support, nutrition, and geriatric syndromes

SUMMARY:
Depending on the YASAM project which was established to home-visit evaluate community-dwelling older adults (80 years of age and over), we aimed to determine the prevalence (prevalence) of geriatric syndromes (dependence, frailty, malnutrition, depression, dementia, comorbidity burden, polypharmacy) in these individuals and to determine possible changes in the follow-up of the patients during the 2-year follow-up period. (HEAVEN trial)

DETAILED DESCRIPTION:
Individuals over the age of 80 who will participate in the YASAM project will first be informed by phone and their appointments will be made. Subsequently, a home visit will be conducted after obtaining verbal and written consent from the patients and their relatives.

The chronic diseases and medications of the patients will be questioned and controlled from the electronic data set. To determine the level of frailty and dependency, the Katz, Lawton-Brody, and Clinical Frailty scales will be filled in, respectively, by the previously trained health personnel, by interviewing their relatives. Mini-Cog, Mini Mental Status Assessment, Mini Nutrition Assessment, and Geriatric Depression (Yesavage) Assessments will be planned. According to dependency status, individuals will be re-evaluated in the 1st or 2nd month. If the patients are fully independent, control follow-up is planned in the 3rd month. Written file records will be created by obtaining the consent of the patients and their relatives at each patient visit. Each team will be responsible for the follow-up of 300 patients. It is planned to include a total of 6000 individuals in the first phase, which is carried out in 20 centers throughout the province of Balıkesir and whose coordination center is Atatürk city hospital. In the follow-ups, it is planned to include the whole cohort consisting of 40 thousand individuals over the age of 80, by increasing the number of teams. The short-term results of the patient's follow-up (1st, 3rd, and 6th-month results), changes in mortality, addiction, frailty level, and changes in nutrition and cognitive functions within the specified period will be evaluated as short-term results. It is aimed to record the long-term outcomes (1st and 2nd year) of the same variables.

Since the whole population will be included in the study, sample size and power analysis were not performed.

ELIGIBILITY:
Inclusion Criteria:

* 80 years and over older adults
* individuals giving verbal and written consent for the YASAM project

Exclusion Criteria:

* <80 years older adults
* those who did not give verbal and written consent for the YASAM project

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: It is planned to include a total of 6000 individuals in the first phase, which is carried out in 20 centers throughout the province of Balıkesir (rural and central area) and whose coordination center is Balikesir Atatürk City Hospital. In the follow-ups, it is planned to include the whole cohort consisting of individuals over the age of 40 thousand 80, by increasing the number of teams.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Short term Healthy Aging status (mortality) | 1-,3-,6- month
  Outcomes were evaluated according to the national electronic database.
Short term Healthy Aging status (changes dependency ) | 1-,3-,6- month
  Outcomes were evaluated according to the specific test Katz scales the 1 is minimum and 6 is maximum value for scale, and higher scores mean a better outcome, higher scores mean a better outcome for dependency)
Short term Healthy Aging status (changes in frailty level) | 1-,3-,6- month
  Outcomes were evaluated according to the specific test (Fraility via Clinical fraility scales the 1 is minimum and 9 is maximum value for scale, and higher scores mean a worse outcome).
Short term Healthy Aging status (changes in nutrition) | 1-,3-,6- month
  Outcomes were evaluated according to the specific test (MNA scale for nutritional status the 0 is minimum and 14 is maximum value for scale, and higher scores mean a better outcome).
Short term Healthy Aging status (changes in cognitive functions) | 1-,3-,6- month
  Outcomes were evaluated according to the specific test (cognitive functions with MMSE scale, the 0 is minimum and 30 is maximum value for scale, and higher scores mean a better outcome)
Short term Healthy Aging status (changes in mood) | 1-,3-,6- month
  Outcomes were evaluated according to the specific test (Outcomes were evaluated according to the specific test ( Yesavage for Depression status the 0 is minimum and 15 is maximum value for scale, and higher scores mean a worse outcome)
Short term Healthy Aging status (changes in mobility status) | 1-,3-,6- month
  Outcomes were evaluated according to the specific test (Chair stand test higher scores (>13,5 seconds) means a worse outcome for mobility status).
Long term Healthy Aging status (mortality) | 1- and 2- year
  Outcomes were evaluated according to the national electronic database.
Long term Healthy Aging status (changes dependency ) | 1- and 2- year
  Outcomes were evaluated according to the specific test Katz scales the 1 is minimum and 6 is maximum value for scale, and higher scores mean a better outcome, higher scores mean a better outcome for dependency)
Long term Healthy Aging status (changes in frailty level) | 1- and 2- year
  Outcomes were evaluated according to the specific test (Fraility via Clinical fraility scales the 1 is minimum and 9 is maximum value for scale, and higher scores mean a worse outcome.)
Long term Healthy Aging status (changes in nutrition) | 1- and 2- year
  Outcomes were evaluated according to the specific test (MNA scale for nutritional status the 1 is minimum and 14 is maximum value for scale, and higher scores mean a better outcome).
Long term Healthy Aging status (changes in cognitive functions) | 1- and 2- year
  Outcomes were evaluated according to the specific test (cognitive functions with MMSE scale, the 0 is minimum and 30 is maximum value for scale, and higher scores mean a better outcome).
Long term Healthy Aging status (changes in mood) | 1- and 2- year
  Outcomes were evaluated according to the specific test ( Yesavage scale for Depression status the 0 is minimum and 15 is maximum value for scale, and higher scores mean a worse outcome).
Long term Healthy Aging status (changes in mobility status) | 1- and 2- year
  Outcomes were evaluated according to the specific test (Outcomes were evaluated according to the specific test (Chair stand test higher scores (>13,5 seconds) means a worse outcome for mobility status).

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Katipoglu, Study Director — Gulhane Training and Research Hospital
Locations (1):
- Balikesir Ataturk City Hospital, Balıkesir, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Katipoglu B, Kocyigit SE, Ergun U, Kocak AO, Aydeniz O, Mert I, Keskin SK. A Community-Based Integrated Healthy Aging Program at a Tertiary Hospital (YASAM) for the Oldest Old Participants May have the Potential to Reduce Emergency Admission: Preliminary Evidence from a Pre-Post-Intervention Study. J Emerg Med. 2025 May;72:112-120. doi: 10.1016/j.jemermed.2024.12.009. Epub 2024 Dec 31. PMID 40316458
- [Derived] Katipoglu B, Kocyigit SE. Impact of geriatric syndrome burden on healthcare services utilization and mortality among community-dwelling older adults: is it still too late to do something? Eur Geriatr Med. 2025 Jun;16(3):1055-1061. doi: 10.1007/s41999-025-01189-w. Epub 2025 Mar 22. PMID 40120075